CLINICAL TRIAL: NCT01087060
Title: Does Hounsfield Unit (HU) Predict the Detection of Cystic Renal Malignancy of Complicated Renal Cysts?
Brief Title: Detection of Renal Malignancy of Complicated Renal Cysts
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Other Study IDs: Bosniak
Record Dates: First submitted 2010-03-10; First posted 2010-03-15 (Estimated); Last update posted 2010-03-15 (Estimated); Status verified 2010-03

CONDITIONS: Kidney Neoplasm; Cysts; Carcinoma, Renal Cell
MeSH Terms: conditions — Kidney Neoplasms; Cysts; Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- cysts surgically removed
  Interventions: Procedure: partial or radical nephrectomy
- cysts under surveillance

INTERVENTIONS:
Procedure: partial or radical nephrectomy
  Groups: cysts surgically removed

SUMMARY:
The aim of this study was to show additional diagnostic criteria of computed tomography (CT) scan to diagnose and predict the detection and recurrence of cystic renal cell carcinoma in the patients with complicated renal cysts. Furthermore, we would demonstrate the relationship between complicated renal cysts diagnosed by Bosniak system and some parameters of pathological results. The analysis about detection time of renal malignancy would help determine the practical guidelines of follow-up plan for complicated renal cysts.

DETAILED DESCRIPTION:
Even though there have been many trials and errors to enhance the diagnostic accuracy of CT scans for complicated cysts, the trial to obtain the enhanced accuracy using CT scan would be still valuable, when we consider its widespread use. A previous study demonstrated that the enhancement of HU with intravenous administration of contrast material on CT scan by 15 HU would be "almost always indicative of a pathologic process although not always a malignancy", another study showed the cut-off as 42 or 47 HU gap would be helpful in the prediction of renal malignancy.

ELIGIBILITY:
Inclusion Criteria:

* All patients who were diagnosed as renal cysts
* available serial follow-up data of CT scan
* all CT imaging included non-enhanced (NEP), corticomedullary (CMP), and early excretory phase (EEP) scans. The scan delay times should range from 30 to 40 seconds for CMP scans and from 120 to 180 seconds for EEP scans.

Exclusion Criteria:

* cases diagnosed by only US/MR
* no serial CT images
* cysts of autosomal dominant adult polycystic kidney disease
* cysts less than 1cm in diameter (difficult to evaluate accurately)
* follow-up period less than 1 yr in the patients who had no surgery

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All 2,992 patients who were diagnosed as renal cysts in this institute
Sampling Method: Probability Sample
Enrollment: 269 (Actual)
Dates: Start 1997-01; Primary Completion 2008-03 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
additional diagnostic criteria of CT to diagnose and predict the detection and recurrence of cystic RCC in the patients with complicated renal cysts
  First, the primary outcomes is to determine cut-off values of maximal HU and the maximal gap of HU (HU of early excretory phase minus that of non-enhanced phase in CT scan)to predict the detection of renal malignancy. Some clinical factors (age, height, body weight, etc) were also included in the analysis.
  Second, the above-mentioned factors were included in the analysis of risk factors for recurrence of complicated renal cysts to determine the cut-off values.

SECONDARY OUTCOMES:
informative to determine the time of operation and which is better for a patient with a complicated cyst between partial or radical nephrectomy
  The cut-off values would show a guideline to determine the time of operation for a patient with complicated renal cysts, namely, the nephrectomy should be performed earlier if the patient is included in the high-risk group. Furthermore, the cut-off value would be helpful in the determination in what operation would be proper to the patient. A partial nephrectomy would be more beneficial to every patient than radical nephrectomy, however, if the patient is in the high-risk group for early recurrence, the patient should undergo 'radical' nephrectomy first for complicated renal cysts.

CONTACTS AND LOCATIONS:
Overall Officials: Cheol Kwak, M.D.,Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Result] Song C, Min GE, Song K, Kim JK, Hong B, Kim CS, Ahn H. Differential diagnosis of complex cystic renal mass using multiphase computerized tomography. J Urol. 2009 Jun;181(6):2446-50. doi: 10.1016/j.juro.2009.01.111. Epub 2009 Apr 17. PMID 19375094